CLINICAL TRIAL: NCT02876770
Title: Nocturnal Melatonin Ingestion Ameliorates Short Term Maximal Performances on the Following Day
Brief Title: Melatonin Supplementation and Performance
Acronym: MSP
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: kais (Other)
Responsible Party: Sponsor-Investigator, kais, Doctor, University of Sfax
Organization: University of Sfax (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CNMSS1
Record Dates: First submitted 2016-08-02; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity

ARMS (2):
- Melatonin (Experimental)
  Interventions: Dietary Supplement: Experimental: Melatonin
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Experimental: Melatonin — Our protocol was composed of three experimental sessions. During each testing session, participants were requested to attend the laboratory at 20:00h where they ingested a standardized light meal. Melatonin (5 mg or 8 mg) or placebo were ingested in capsule in the evening at 21:00h in a double-blind randomized design
  Arms: Melatonin
Dietary Supplement: Placebo — In a double-blind randomized design, participants have taken placebo supplementation in one of the three experimental sessions
  Arms: Placebo

SUMMARY:
The present study aimed to evaluate the possible effect of nocturnal melatonin ingestion upon short-term performances, on the following morning. Twelve soccer players from a Tunisian squad (22.9 ±1.3 years, 1.80±0.05 m, and 72.0±8.8 kg) were volunteered to perform three testing sessions, with one test session per day. During each session, MEL (5mg) , MEL (8mg) or placebo were ingested, in a randomized order, before nocturnal sleep. The next morning (08:00h), participants performed the following psycho-cognitive and physical tests: Hooper's index, reaction time, vigilance, handgrip strength , squat jump , modified agility test , Wingate anaerobic test (peak power , mean power and fatigue index ). Rating of perceived exertion was recorded immediately after the WanT, and blood lactate measures were taken after 3min of recovery. Blood glucose was measured before and 3 min after the Wingate test.

ELIGIBILITY:
Inclusion Criteria:

The participants were recruited based on the following criteria: (i) paticipants must be trained at 4-6 days per week for an average of 2 h daily and (ii) they must have at least 8 years of training experience

Exclusion Criteria:

* Subjects were excluded from the study if they present one of the following criteria : heart failure, antioxidant supplementation within 3 months before the study, lower-limb injuries

Ages: 20 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Hooper's index score | At 07:30 am in the following day of the supplementation
  Hooper's index score was measured using a specific questionnaire
handgrip strength (in Kg) | At 07:30 am in the following day of the supplementation
  handgrip strength was measured using a calibrated hand dynamometer.
Blood lactate (µmol/l) | Blood lactate was measured only 3 minutes after physical testing in the following day of the supplementation
  Lactate level was measured using Lactate Pro instrument.
reaction time (in secondes) | At 07:30 am in the following day of the supplementation
  Reaction time was measured using an electronic timing device.
vigilance score | At 07:30 am in the following day of the supplementation
  Vigilance score was measured using a specific questionnaire
squat jump (in centimeters) | At 07:30 am in the following day of the supplementation
  Squat jump was assessed using a infrared jump system
agility (in secondes) | At 07:30 am in the following day of the supplementation
  Agility was assessed using an electronic timing system.
anaerobic capacity (In watts) | At 07:30 am in the following day of the supplementation
  Anaerobic capacity was assessed using a calibrated friction-loaded cycle ergometer
glucose level (µmol/l) | At 07:30 am in the following day of the supplementation (rest condition) and 3 minutes after physical testing in each experimental session
  Glucose level was assessed using a glucometer
Rating of perceived exertion score | Rating of perceived exertion score was measured 3 minutes after physical testing in the following day of the supplementation
  Rating of perceived exertion score was measured using a specific questionnaire